CLINICAL TRIAL: NCT06998719
Title: A Phase II, Interventional Study of Neoadjuvant Durvalumab and Platinum-based Chemotherapy, Followed by Surgery and Adjuvant Durvalumab or Chemoradiotherapy and Consolidation Durvalumab, in Borderline Resectable Stage III NSCLC (ACCESS)
Brief Title: Neoadjuvant Durvalumab and Chemotherapy Followed by Surgery/CRT and Durvalumab in Borderline Resectable Stage III NSCLC
Acronym: ACCESS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bi Nan (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Bi Nan, Chief physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5253
Record Dates: First submitted 2025-04-21; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer Stage III; Borderline Resectable Carcinoma
Keywords: Neoadjuvant therapy; Non-small Cell Lung Cancer; Borderline Resectable Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Surgical Procedures, Operative; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Surgery) (Experimental): After 2 cycles of neoadjuvant durvalumab (1500 mg) + chemotherapy, multidisciplinary team (MDT)-determined participants with resectable tumor (according to MDT re-assessment) will receive a further 1-2 cycles of neoadjuvant durvalumab + chemotherapy followed by surgery. Participants should only go onto surgical resection if the MDT evaluation indicates that an R0 resection is feasible.
  After surgery, patients will then go on to receive adjuvant durvalumab 1500 mg q4w until recurrence or up to one year (maximum 12 cycles) unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Interventions: Drug: Durvalumab
- Cohort 2 (CRT) (Active Comparator): Participants with unresectable tumor (according to MDT re-assessment) will receive CRT. Participants will receive platinum-based chemotherapy for a maximum of 2 cycles. Radiotherapy at a dose of 5 fractions/week for ~6 weeks (± 3 days) (total 60 Gy± 10%) can be given sequentially or concurrently with chemotherapy.
  After CRT, patients will receive consolidation durvalumab 1500 mg q4w until disease progression or up to one year (maximum 12 cycles) unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Neoadjuvant durvalumab (MEDI 4736)and platinum-based chemotherapy, followed by either surgery and adjuvant durvalumab or CRT and consolidation durvalumab, in borderline resectable stage III NSCLC
  Other Names: Surgery; Chemoradiotherapy (CRT)

SUMMARY:
A Phase II, interventional study of neoadjuvant durvalumab (MEDI 4736) and platinum-based Chemotherapy, followed by either surgery and adjuvant durvalumab or chemoradiotherapy (CRT) and consolidation durvalumab, in participants with borderline resectable stage III Non-small Cell Lung Cancer (NSCLC) (ACCESS)

DETAILED DESCRIPTION:
This is a multicenter, Phase II, Chinese study assessing the efficacy and safety of neoadjuvant durvalumab and platinum-based Chemotherapy, given intravenously, followed by either surgery and adjuvant durvalumab or definitive CRT and consolidation durvalumab in participants with borderline resectable stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participant must be ≥ 18 years, at the time of screening. 2. Histologically or cytologically documented NSCLC. 3. Deemed borderline resectable at baseline, confirmed by MDT evaluation at diagnosis.

  4. Previously untreated and pathologically confirmed stage III (according to Version 8 of the IASLC Staging Manual in Thoracic Oncology2016)
  1. Nodal status should be investigated with whole body FDG-PET, plus contrast-enhanced computed tomography, and it is optional and decided by investigator that nodal status be proven by biopsy via endobronchial ultrasound, mediastinoscopy, or thoracoscopy.
  2. Mandatory brain MRI with IV contrast, if not available, it is mandatory to take brain computed tomography with IV contrast at the time of staging.

     5. WHO or ECOG performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline or day of first dose.

     6. Participants must have been confirmed as EGFR/ALK wild type via an appropriately validated local test. Participants with known sensitising EGFR mutations or ALK rearrangements are excluded from the study.

     7. At least one lesion not previously irradiated that qualifies as a RECIST 1.1 TL at baseline and can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes, which must have short axis ≥ 15 mm) with computed tomography or MRI and is suitable for accurate repeated measurements.

     8. Adequate organ and bone marrow function as follows:
* Haemoglobin ≥ 9.0 g/dL.
* Absolute neutrophil count ≥ 1.5 × 109/L.
* Platelet count ≥ 100×109/L.
* Serum bilirubin ≤ 1.5×the ULN or ≤ 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinaemia).
* Alanine aminotransferase and AST ≤ 2.5×ULN.
* Calculated CrCL > 40 mL/min as determined by Cockcroft Gault (using actual body weight).

Males:

CrCL (mL/min) = Weight (kg) × (140 - Age) 72 × serum creatinine (mg/dL)

Females:

CrCL (mL/min) = Weight (kg) × (140 - Age) × 0.85 72 × serum creatinine (mg/dL) 9. Minimum life expectancy of 12 weeks. 10. The participant should be deemed to have adequate cardiac and lung function, according to a multidisciplinary assessment. A pre- or post-bronchodilator FEV1 of 1.0 L and >40% post-operative predicted value. Use of these cut-off values to assess candidacy for resection on pre-treatment risk assessment. (Surgical Eligible) 11. Minimum body weight of 30 kg. 12. Negative pregnancy test (serum) for FOCBP for female. 13. Male participants who intend to be sexually active with a female partner of child-bearing potential must be surgically sterile or using an acceptable method of contraception from the time of screening, while receiving study intervention, SoC Chemotherapy or CRT, and for 90 days after the last dose of durvalumab and for periods specified in the local prescribing information/SmPC relating to contraception and the time limit for such precautions for SoC agents to prevent pregnancy in a partner. Male participants must not donate or bank sperm during this same time period.

14. Female participants must be for 1 year or more post-menopausal, surgically sterile, or using at least one highly effective method of contraception: a highly effective method of contraception is defined Non-hormonal

* Total sexual abstinence (evaluate in relation to the duration of the clinical study and the preferred and usual lifestyle choice of the participant)
* Vasectomised sexual partner (with participant assurance that partner received post-vasectomy confirmation of azoospermia)
* Tubal occlusion Intrauterine device (provided coils are copper banded) Hormonal
* Implants: Etonogestrel-releasing implants (e.g. Implanon® or Norplant®)
* Intravaginal devices: Ethinylestradiol/etonogestrel-releasing intravaginal devices (e.g. NuvaRing®)
* Injection: Medroxyprogesterone injection (e.g. Depo-Provera®)a
* Combined Pill: Normal and low dose combined oral contraceptive pill
* Patch: Norelgestromin/ethinylestradiol-releasing transdermal system (e.g. Ortho Evra®)
* Mini pill: Progesterone based oral contraceptive pill using desogestrel: Cerazette® is currently the only highly effective progesterone-based Levonorgestrel-releasing intrauterine system (e.g., Mirena®)

  1. Females < 50 years old are considered post-menopausal if they have been amenorrhoeic for 12 months or more prior to enrolment following cessation of exogenous hormonal treatment and follicle-stimulating hormone (FSH) levels in the post-menopausal range.
  2. Females ≥ 50 years old are considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment, or had radiation-induced menopause with last menses > 1 year ago, or had chemotherapy-induced menopause with last menses > 1 year ago.
  3. Female participants of child-bearing potential must agree to use at least one highly effective method of birth control (see Appendix G for complete list of highly effective birth control methods). They should have been stable on their chosen method of birth control for a minimum of 3 months prior to enrollment (screening), while receiving study intervention, SoC Chemotherapy or CRT, and for 90 days after the last dose of durvalumab and for periods specified in the local prescribing information/SmPC relating to contraception and the time limit for such precautions for SoC agents. Cessation of birth control after this point should be discussed with a responsible physician.
  4. Non-sterilised male partners of a female participant of child-bearing potential must use a male condom plus spermicide (condom alone in countries where spermicides are not approved) from the time of screening their female partner, while their female partner is receiving study intervention, SoC Chemotherapy or CRT, and for 90 days after the last dose of durvalumab and for periods specified in the local prescribing information/SmPC relating to contraception and the time limit for such precautions for SoC agents.
  5. Periodic abstinence, as well as the rhythm and withdrawal methods are not acceptable methods of birth control..

     15. Capable of giving signed informed consent as described in Appendix which includes compliance with the requirements and restrictions listed in the ICF and in this CSP.

     16. Provision of signed and dated written Optional Genetic Research Information informed consent prior to collection of samples for optional genetic research that supports the Genomic Initiative.

     17. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

     Exclusion Criteria:
     1. Existence of more than one primary tumor, such as: mixed small cell and NSCLC histology; synchronous or metachronous tumors that could represent distinct primary tumors.
     2. History of another primary malignancy except for malignancy treated with curative-intent with no known active disease ≥ 5 years before the first dose of study intervention and of low potential risk for recurrence, basal cell carcinoma of the skin, squamous cell carcinoma of the skin or lentigo maligna that has undergone potentially curative therapy or adequately treated carcinoma in situ without evidence of disease.
     3. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis or Crohn's disease], systemic lupus erythematosus, sarcoidosis, granulomatosis with polyangiitis, Graves ' disease, rheumatoid arthritis, hypophysitis, uveitis, autoimmune pneumonitis, and autoimmune myocarditis). The following are exceptions to this criterion:

        - Participants with vitiligo or alopecia.

        - Participants with hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement.

        - Any chronic skin condition that does not require systemic therapy.

        - Participants without active disease in the last 5 years may be included but only after consultation with the Study Clinical Lead.

        - Participants with coeliac disease controlled by diet alone.
     4. Known active hepatitis infection, positive HCV antibody, HBsAg or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti-HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Participants co-infected with HBV and HCV, or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti-HBcAb with detectable HBV DNA); AND

        * HCV positive (presence of anti-HCV antibodies); OR
        * HDV positive (presence of anti-HDV antibodies).
     5. Known to have tested positive for HIV (positive HIV 1 or 2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice).
     6. History of active primary immunodeficiency.
     7. Investigator judgement of one or more of the following:

        * Mean resting corrected QT interval > 470 ms, obtained from triplicate ECGs performed at screening.
        * History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and cause TdP.
        * Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden cardiac death under 40 years of age in first-degree relatives.
     8. Prior exposure to immune-mediated therapy including, but not limited to, other anti-CTLA-4, anti-PD-1, anti-PD-L1 and anti-PD-L2 antibodies, excluding therapeutic anticancer vaccines.
     9. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

        - Intranasal, inhaled, topical steroids or local steroid injections (eg, intra-articular injection).
        * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
        * Steroids as premedication for hypersensitivity reactions or as an anti-emetic (eg, computed tomography scan premedication).
     10. Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention.
     11. Major surgical procedure or significant traumatic injury within 4 weeks of the first dose of study intervention.
     12. Any medical contraindication to treatment with platinum-based doublet Chemotherapy, as listed in the local labelling.
     13. Previous treatment in the present study or a previous durvalumab clinical study regardless of treatment arm assignment.
     14. Participation in another clinical study with a study intervention administered in the last 4 weeks prior to first dose of durvalumab or concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
     15. Participants with a known hypersensitivity to durvalumab or any excipients of the product(s).
     16. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
     17. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
     18. Female participants who are pregnant or breastfeeding or male or female participants of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy. Specifically, regarding the receipt of SoC chemotherapy or chemoradiotherapy, participants should be willing to follow the local prescribing information relating to contraception, the time limits for such precautions, and any additional restrictions for the agents administered.
     19. Participants with a documented test result confirming the presence of a known EGFR or ALK sensitizing mutation is excluded from the study.
     20. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤28 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator.
     21. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria:

     <!-- -->

     1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.

     22. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.

     (2) History of allogenic organ transplantation. (3) History of leptomeningeal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Resection rate | Through study completion, an average of 1 year.
  To assess the efficacy of neoadjuvant durvalumab + chemotherapy in terms of resection rate in participants with borderline resectable stage III NSCLC.

SECONDARY OUTCOMES:
R0 resection rate. | Through study completion, an average of 1 year.
  To investigate surgical outcomes.R0 resection indicates a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.R0 resection rate =The number of subjects whose lesions were completely removed/the number of subjects who participated in the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No